CLINICAL TRIAL: NCT00869622
Title: Antiepileptic Drugs and Osteoporotic Prevention Trial
Acronym: ADOPT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston VA Research Institute, Inc. (Other)
Collaborators: Procter and Gamble (Industry); Alliance for Better Bone Health (Other); VA Boston Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Antonio Lazzari, Director Osteoporosis Prevention and Treatment Center VABHCS, Boston VA Research Institute, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VABHS IRB#1889
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Results first posted 2015-07-24 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Epilepsy; Bone Loss; Osteoporosis; Fractures
Keywords: osteoporosis; bone mineral density; fracture; antiepileptic drug; seizure; Prevention of bone loss; Prevention of osteoporosis; Prevention of Fractures
MeSH Terms: conditions — Epilepsy; Bone Diseases, Metabolic; Osteoporosis; Fractures, Bone; Seizures | interventions — Risedronic Acid; Calcium; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Risedronate (Active Comparator): Active drug
  Interventions: Drug: Risedronate
- Placebo + Calcium and Vitamin D (Placebo Comparator): All patients both on placebo and active bisphosphonate to receive calcium and vitamin D
  Interventions: Drug: Placebo + Calcium and Vitamin D

INTERVENTIONS:
Drug: Risedronate — 35 mgs/week + calcium and vit d
  Other Names: Actonel
  Arms: Risedronate
Drug: Placebo + Calcium and Vitamin D — sugar pill + calcium 1200mgs/day and vitamin d at least 800IU
  Other Names: Placebo
  Arms: Placebo + Calcium and Vitamin D

SUMMARY:
Study Design: (e.g., Controlled, Double-Blind, Randomized, Parallel):

Randomized, double-blind, placebo controlled of a bisphosphonate in the prevention of bone loss associated with the use of antiepileptic drugs.

DETAILED DESCRIPTION:
The study is planned to last two years. You will be required to make a total of 6 visits to the clinic during this two year study period. At the first visit, 12 months and, approximately 24 months, you will have a bone mineral density test (BMD) of your hip and spine. A BMD is similar to having an x-ray and is a test that measures the amount of bone. This test takes approximately 15 minutes. Radiation exposure during this test is very low. It has been estimated that the total radiation exposure from a bone mineral density measurement is lower than that of a dental x-ray. At each follow up visit an assessment will be made for side effects and whether or not you followed the prescribed treatment.

Initially, information collected will include height, weight, seizure history and seizure medication history, other medical conditions, bone and muscle symptoms you currently have, dietary calcium intake, and exercise. Blood will be drawn at the initial and 5 follow-up visits. The purpose of this is to test your blood for organ function, calcium levels, vitamin D levels and levels of markers that show high bone turnover. Also at each visit your height and weight will be checked and you will be asked questions regarding side effects, adherence to treatment and quality of life.

When you agree to participate, you will be randomized to either risedronate 35mg tablet (Actonel ®) or placebo (a fake pill) to take once a week. Randomization is a process in which you will have an equal chance (like the flip of a coin) to be assigned to either risedronate (Actonel ®) or placebo. A computer program will determine your treatment assignment. Also during the study you will be provided with calcium and vitamin D tablets to take either two or three times each day depending on your dietary calcium intake.

At the first visit you will be assessed for changeable risk factors for osteoporosis. These include smoking, alcohol consumption, and lack of physical activity, poor nutrition and lack of vitamin intake. Also, blood will be drawn to see if you have a low male hormone. If you are found to have low male hormone, you will be referred to your primary care provider. If you have low male hormone levels, you will be eligible to participate in the study if testosterone replacement has been offered to you and you have declined treatment. If you decide to be treated with testosterone you are not eligible to participate in this study. Education will be provided on exercises for bones. If you smoke, you will be counseled on quitting although quitting is not a requirement to participate in the study. If you drink a lot of alcohol you will be counseled on reducing your intake and offered help. Reducing or quitting alcohol is not a requirement for your participation in this study. You can also meet with a registered dietician for nutritional counseling.

ELIGIBILITY:
Inclusion Criteria:

* Male gender
* Epilepsy
* Anti-epileptic drug treatment with phenytoin, or phenobarbital or valproate sodium
* Normal renal function and normal Vitamin D and calcium levels

Exclusion Criteria:

* Female gender
* Organ transplant
* Use of oral glucocorticoids
* Renal insufficiency (eGFR < 30ml/min)
* Severe swallowing disorder
* Severe esophagitis
* Patients taking sodium valproate for reasons other than epilepsy
* Previous treatment with osteoporosis drugs such as bisphosphonates, calcitonin or PTH analog

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2006-06; Primary Completion 2012-10 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio A Lazzari, MD, Principal Investigator — VA Boston HCS; Phillip Dussault, Pharm D, Principal Investigator — VA Boston HCS; Manisha Thakore, MD, Principal Investigator — VA Boston HCS
Locations (1):
- VA Boston Healthcare System, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 80 veterans with epilepsy who were treated with phenobarbital, phenytoin, carbamazepine and sodium valproate.
Pre-assignment Details: 80 epileptic patients who have been on phenytoin, phenobarbital, carbamazepine or sodium divalproex for at least 2 years were enrolled.
Groups:
- Placebo Sugar Pill: All patients both on placebo and active bisphosphonate to receive calcium and vitamin D
  Placebo + calcium and vitamin d: sugar pill + calcium 1200mgs/day and vitamin d at least 800IU
Period: Overall Study
Arm/Group | Risedronate | Placebo Sugar Pill
Started | 40 | 40
Completed | 27 | 26
Not Completed | 13 | 14

BASELINE CHARACTERISTICS:
Groups:
- Risedronate: Active drug participants received calcium and vitamin D supplementation in addition to 35 mgs of risedronate tablet weekly
- Placebo Sugar Pill: Placebo participants received calcium and vitamin D supplementation in addition to a placebo tablet identical to risedronate tablet weekly
- Total: Total of all reporting groups
Arm/Group | Risedronate | Placebo Sugar Pill | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 29 | 50
  >=65 years | 19 | 11 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (13) | 58 (13) | 61 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 40 | 40 | 80
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80
Type of seizures [Number; unit: participants]
  Grand Mal Seizures | 19 | 22 | 41
  Other types of seizures | 21 | 18 | 39
Current Smokers [Number; unit: participants]
  Smokers | 29 | 28 | 57
  Non Smokers | 11 | 12 | 23
Baseline Vitamin D Level [Mean (Standard Deviation); unit: ng/ml] | 29.1 (19) | 29.3 (16) | 29.2 (17.5)
Previous Vertebral Fractures [Number; unit: participants]
  Previous vertebral fractures | 15 | 9 | 24
  No veterbral fractures | 25 | 31 | 56

OUTCOME MEASURES:

1. Primary Outcome: Changes in Bone Mineral Density
Description: Patients with a T-Score of > -2.5 were randomized into two possible arms. A bisphosphonate group received 35mg risedronate weekly while another group received an identical placebo tablet weekly. Both groups received supplemental calcium and vitamin D.
  Enrolled patients had bone density measurements of bilateral proximal femur, A-P lumbar spine, total body, forearm and L-P spine. All measurements were performed on a GE Lunar Bone Densitometer (iDXA) instrument. Measurements of 25-hydroxy vitamin D, NTX , serum calcium and blood chemistries occurred at scheduled intervals.
Time Frame: 2 years
Population: The study design involved 80 veterans with epilepsy who were treated with phenobarbital, phenytoin, carbamazepine and sodium valproate. This is a prospective study in which 80 patients who have been on phenytoin, phenobarbital, carbamazepine or sodium divalproex for at least 2 years were enrolled.
Measure: Mean (Standard Deviation); unit: g/cm2
Arm/Group | Risedronate | Placebo Sugar Pill
Number analyzed (Participants) | 27 | 26
g/cm2
  Bilateral Proximal Femora | 1.025 (0.111) | 0.999 (0.174)
  L1-L4 AP Spine | 1.332 (0.111) | 1.245 (0.154)
  Total Body BMD | 1.205 (0.096) | 1.192 (0.127)

2. Secondary Outcome: Vertebral Fractures
Time Frame: 2 years
Measure: Number; unit: Vertebral Fractures
Arm/Group | Risedronate | Placebo + Calcium and Vitamin D
Number analyzed (Participants) | 27 | 26
Vertebral Fractures | 0 | 5
Statistical Analysis 1: Comparison: Risedronate vs Placebo + Calcium and Vitamin D; Test type: Superiority or Other; p = 0.0229, Fisher Exact

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Risedronate | Placebo Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No